CLINICAL TRIAL: NCT05977517
Title: Sleep, Learning and Wellbeing in NUS Undergraduates: The NUS1000 Study
Acronym: NUS1000
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Michael W.L. Chee, Professor, National University of Singapore
Other Study IDs: NUS1000
Record Dates: First submitted 2023-06-27; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Sleep; Well-Being, Psychological
MeSH Terms: conditions — Psychological Well-Being | interventions — Sleep

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Sleep and well-being tracking — This study will track sleep, learning and wellbeing of 500 freshmen under free-living conditions for 20 weeks

SUMMARY:
NUS1000 is a large scale freshman-year study of undergraduate sleep, well-being and learning patterns that has unique key features: (1) continuous objective multi-dimensional data gathered with passive sensing of sleep and stress over a semester, (2) utilisation of Learning Management System-based outcome data as a marker of study behaviour and academic achievement. The goal is to gather information that can be used to improve student sleep, mental wellbeing and performance.

DETAILED DESCRIPTION:
The first year in university can be a challenging experience for undergraduates who must learn to cope with learning in an unfamiliar environment, form new relationships, live away from home and/or might have to manage personal finances for the first time. These academic, social, and personal demands can result in significant stress, affecting sleep, learning and mental/emotional wellbeing. Characterizing and understanding the time-course and inter-relationship of these demands and their consequences is crucial for making science-based improvements to a student's university experience. To this end, the investigators will longitudinally evaluate sleep, learning and wellbeing in ~1000 first-year students as they adapt to university life to understand how these behaviours fluctuate and interact throughout the academic term.

ELIGIBILITY:
Inclusion Criteria:

* NUS first-year students with smartphones operating on Android 8.0 and up, or iOS 14.0 or later

Exclusion Criteria:

Participants will be required to :

1. Have their sleep and physical activity rhythms will be recorded via wearable sensors, while they continue daily life as usual.
2. Complete periodic questionnaires, short daily surveys and daily audio diaries on their smartphones.
3. Agree to interactions with their smartphones and as well as grades tracked. Participants who do not agree to have these measures recorded will not be eligible for the study.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: NUS Freshmen students
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Change in sleep duration and timing from the start to the end of the semester | 20 weeks
  The Oura ring is a sleep-tracking device worn on the finger. During the study, participants will need to sync their devices to a mobile app.
Change from baseline sleep habits from the start to the end of the semester | Week 1-2, Week 8-9, and Week 17-18
  Participants will also be required to complete a set of sleep questionnaires probing sleep habits (bedtime, wake time, time taken to fall asleep, etc.)
Change in daily well-being from the start to the end of the semester | 20 weeks
  Participants will be prompted to fill in brief questions on daily well-being. At the end of each assessment, participants will be required to record an audio clip of their day, without any personal identifiers, for mood/sentiment analysis.
Change from baseline well being from the start to the end of the semester | Week 1-2, Week 8-9, and Week 17-18
  Participants will also be required to complete a set of well-being questionnaires (e.g., feelings of connectedness or isolation, levels of stress, etc.)
Change in learning outcomes from the start to the end of the semester | 20 weeks
  Grades from quiz/assignments for each module will be collected.
Change in learning patterns from the start to the end of the semester | 20 weeks
  Student interactions with the LMS-system will be collected, such as the number of page/file views.
Change in mood from the start to the end of the semester | 20 weeks
  At the end of each day, participants will be required to record an audio clip of their day, without any personal identifiers, for mood analysis.
Change in time-use patterns from the start to the end of the semester | Week 1-2, Week 8-9, and Week 17-18
  Participants will be asked to fill out a time-use diary over three 2-week periods throughout the semester, indicating the activities they engaged in over the past day
Change in smartphone touchscreen interaction patterns from the start to the end of the semester | 20 weeks
  Phone taps will be tracked automatically through an EU-GDPR (the European Union's stringent privacy regulation) compliant smartphone app (QuantActions). This application logs human-smartphone screen interactions during regular use by logging a location-specific timestamp for each screen contact.

SECONDARY OUTCOMES:
Change in movement patterns from the start to the end of the semester | 20 weeks
  The investigator's in-house smartphone app (Z4IP) will extract movement patterns from location data that will only be kept on the participant's phone up to 96 hours for these computations. The extracted movement patterns (and not geographical locations) will then be uploaded to secure servers, tagged to subject IDs without any personal identifiers, i.e., names and emails will not be linked to their movement patterns. As this component is optional, participants will be asked to indicate if they would like to opt-in at the informed consent stage.

IPD SHARING:
Plan to Share IPD: Undecided